CLINICAL TRIAL: NCT01286311
Title: Tailored Communication to Reduce Cardiovascular Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Stephen Persell, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Reducing CV Risk; K08HS015647 (AHRQ)
Record Dates: First submitted 2011-01-27; First posted 2011-01-31 (Estimated); Results first posted 2015-02-09 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-01

CONDITIONS: Hypercholesterolemia; Coronary Artery Disease; Dyslipidemia; Hypertension
Keywords: Health Education; Health Knowledge, Attitudes, Practice; Hypolipidemic Agents/therapeutic use; Patient Education as Topic
MeSH Terms: conditions — Hypercholesterolemia; Coronary Artery Disease; Dyslipidemias; Hypertension; Health Education; Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Direct-to-patient tailored cardiovascular risk message system (Experimental): Eligible patients cared for by physicians randomized to the active intervention group will be mailed a tailored cardiovascular risk message.
  Interventions: Behavioral: Direct-to-patient tailored cardiovascular risk message system
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Direct-to-patient tailored cardiovascular risk message system — Patient informational mailings
  Arms: Direct-to-patient tailored cardiovascular risk message system

SUMMARY:
The primary goal of the trial is to test the feasibility and efficacy of a cardiovascular disease quality improvement system that couples EMR-based patient identification with individually tailored patient messages. The study will test the hypothesis that that a tailored patient-directed approach to cardiovascular risk reduction integrated into patients' primary care delivery site will improve control of elevated low-density lipoprotein cholesterol and other card iac risk factors more than routine care alone for patients at intermediate or high risk for cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 to 79 years
* medication list does not include an active lipid lowering medication
* the patient does not have a diagnosis in the past medical history, active problem list or past visit encounter of coronary heart disease, heart failure, stroke, diabetes mellitus, or peripheral arterial disease
* the patient has an enrolled study physician recorded as his/her primary care physician
* the patient has an LDL cholesterol that meets one or more of the criteria listed below.

LDL cholesterol >= 130 mg/dl and estimated Framingham Risk Score 10-20% LDL cholesterol >= 100 mg/dl and estimated Framingham Risk Score >20% LDL cholesterol >= 160 mg/dl and estimated Framingham Risk Score 5% to <10%.

Exclusion Criteria:

* Age <40 or >79 years
* medication list includes an active lipid lowering medication
* the patient hase a diagnosis in the past medical history, active problem list or past visit encounter of coronary heart disease, heart failure, stroke, diabetes mellitus, or peripheral arterial disease
* the patient does not have an enrolled study physician recorded as his/her primary care physician
* the patient does not have an LDL cholesterol that meets one or more of the criteria listed below.

LDL cholesterol >= 130 mg/dl and estimated Framingham Risk Score 10-20% LDL cholesterol >= 100 mg/dl and estimated Framingham Risk Score >20% LDL cholesterol >= 160 mg/dl and estimated Framingham Risk Score 5% to <10%.

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 464 (Actual)
Dates: Start 2011-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Persell, MD, MPH, Principal Investigator — Northwestern University Division of General Internal Medicine, Feinberg School of Medicine and Institute for Healthcare Studies
Locations (1):
- Northwestern Medical Faculty Foundation General Internal Medicine Ambulatory Clinic, Chicago, Illinois, United States

REFERENCES:
- [Derived] Persell SD, Lloyd-Jones DM, Friesema EM, Cooper AJ, Baker DW. Electronic health record-based patient identification and individualized mailed outreach for primary cardiovascular disease prevention: a cluster randomized trial. J Gen Intern Med. 2013 Apr;28(4):554-60. doi: 10.1007/s11606-012-2268-1. Epub 2012 Nov 11. PMID 23143672

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Physicians were recruited at their clinic offices in January 2011. They provided written informed consent to be randomized and to have study staff mail risk messages directly to patients on their behalf if they were randomized to the intervention. Patients were included with a waiver of consent.
Groups:
- Control: Eligible patients cared for by physicians randomized to the control group will receive usual care. After 9 months, control group physicians were provided with lists of their eligible patients and their risk scores.
Period: Overall Study
Arm/Group | Direct-to-patient Tailored Cardiovascular Risk Message System | Control
Started | 232 (218 patients (of the 14 physician randomized to the intervention) started the study.) | 232 (217 patients (of the 15 physician randomized to the intervention) started the study.)
Completed | 218 (204 patients (of the 14 physician randomized to the intervention) completed the study.) | 232 (217 patients (of the 15 physician randomized to the intervention) completed the study.)
Not Completed | 14 | 0
Not completed — Physician did not want outreach sent | 14 | 0

BASELINE CHARACTERISTICS:
Population: 218 patients (of the 14 physician randomized to the intervention) and 217 patients (of the 15 physician randomized to the intervention) participated in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Direct-to-patient Tailored Cardiovascular Risk Message System | Control | Total
Number analyzed (Participants) | 232 | 232 | 464
Age, Categorical [Number; unit: patient participants] — Physicians were not enrolled according to age criteria, and are therefore not included above.
  patient participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 137 | 147 | 284
    >=65 years | 81 | 70 | 151
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (9.4) | 60.1 (9.2) | 60.7 (9.4)
Gender [Number; unit: participants] — Physicians were not enrolled according to gender criteria, and are therefore not included above.
  participants
    Female | 49 | 50 | 99
    Male | 169 | 167 | 336
Region of Enrollment [Number; unit: participants]
  United States | 232 | 232 | 464

OUTCOME MEASURES:

1. Primary Outcome: Comparative Outcomes: Intervention Group LDL Reduction Compared to Control Group LDL Reduction
Description: Significant LDL cholesterol reduction at 9 months Definition: Percentage of patients with LDL-C repeated and which is at least 30 mg/dl lower than baseline
Time Frame: 9 months
Measure: Number; unit: % of patients with major LDL reduction
Groups:
- Control: Eligible patients cared for by physicians randomized to the control group will receive usual care.
Arm/Group | Direct-to-patient Tailored Cardiovascular Risk Message System | Control
Number analyzed (Participants) | 218 | 217
% of patients with major LDL reduction | 11.0 | 11.1
Statistical Analysis 1: Comparison: Direct-to-patient Tailored Cardiovascular Risk Message System vs Control; Test type: Superiority or Other; p = 0.99, Generalized Logistic Regression; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.54 to 1.86]

2. Secondary Outcome: Frequency of Clinical Encounters
Description: This will measure the difference in frequency of clinical encounters in the electronic medical record.
Time Frame: 9 months
Measure: Number; unit: % of patients with any office visit
Arm/Group | Direct-to-patient Tailored Cardiovascular Risk Message System | Control
Number analyzed (Participants) | 218 | 217
% of patients with any office visit | 61.9 [0 to 2] | 56.7 [0 to 1]
Statistical Analysis 1: Comparison: Direct-to-patient Tailored Cardiovascular Risk Message System vs Control; Test type: Superiority or Other; p = 0.27, Generalized Logistic Regression; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.84 to 1.85]

3. Secondary Outcome: Medication Prescriptions for Dyslipidemia
Description: This will look at whether lipid lowering medications (LLM) were prescribed for dyslipidemia.
Time Frame: 9 months
Measure: Number; unit: % of patients with New Rx for LLM
Arm/Group | Direct-to-patient Tailored Cardiovascular Risk Message System | Control
Number analyzed (Participants) | 218 | 217
% of patients with New Rx for LLM | 11.9 | 6.0
Statistical Analysis 1: Comparison: Direct-to-patient Tailored Cardiovascular Risk Message System vs Control; Test type: Superiority or Other; p = 0.038, Generalized Logistic Regression; Odds Ratio (OR) = 2.13, 95% CI 2-sided [1.05 to 4.32]

4. Secondary Outcome: Percentage of Patients With Uncontrolled Hypertension Who Had an Increase in the Number of Antihypertensive Medication Drug Classes Prescribed
Description: This will measure the percentage of participants who had uncontrolled hypertension at baseline who had an increase in the number of antihypertensive medication drug classes prescribed within 9 months.
Time Frame: 9 months
Population: Among patients with uncontrolled hypertension, 76 of the 218 in the intervention arm and 85 of 217 in the control arm were included.
Measure: Number; unit: percentage of participants
Arm/Group | Direct-to-patient Tailored Cardiovascular Risk Message System | Control
Number analyzed (Participants) | 76 | 85
percentage of participants | 11.8 | 4.7
Statistical Analysis 1: Comparison: Direct-to-patient Tailored Cardiovascular Risk Message System vs Control; Test type: Superiority or Other; p = 0.13, Generalized Logistic Regression; Odds Ratio (OR) = 2.72, 95% CI 2-sided [0.73 to 10.1]

5. Secondary Outcome: Presence of an Aspirin Prescription
Description: This will measure the presence of an aspirin prescriptions on the medication list in the electronic medical record.
Time Frame: 9 months
Population: 38 patients in the intervention arm and 50 patients in the control arm had aspirin listed in their medication list in the electronic medical record as the start of the study therefore they were excluded from this analysis.
Measure: Number; unit: % patients w/aspirin now on med list
Arm/Group | Direct-to-patient Tailored Cardiovascular Risk Message System | Control
Number analyzed (Participants) | 180 | 167
% patients w/aspirin now on med list | 3.9 | 1.8
Statistical Analysis 1: Comparison: Direct-to-patient Tailored Cardiovascular Risk Message System vs Control; Test type: Superiority or Other; p = 0.30, Generalized Logistic Regression; Odds Ratio (OR) = 2.18, 95% CI 2-sided [0.50 to 9.5]

ADVERSE EVENTS:
Description: Serious and/or other [non-serious] adverse events were not collected/addressed. As a result, no participants were at risk.
Arm/Group | Direct-to-patient Tailored Cardiovascular Risk Message System | Control
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No